CLINICAL TRIAL: NCT02282761
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Antipsychotic Efficacy of ITI-007 in Patients With Schizophrenia
Brief Title: A Trial to Assess the Antipsychotic Efficacy of ITI-007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-301
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lumateperone 28 mg (ITI-007 40 mg Tosylate) (Experimental): Lumateperone 28 mg (ITI-007 40 mg Tosylate) administered orally as formulated capsules once daily for 28 days
  Interventions: Drug: ITI-007
- Lumateperone 42 mg (ITI-007 60 mg Tosylate) (Experimental): Lumateperone 42 mg (ITI-007 60 mg Tosylate) administered orally as formulated capsules once daily for 28 days
  Interventions: Drug: ITI-007
- Placebo (Placebo Comparator): Placebo administered orally as formulated capsules once daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ITI-007
  Arms: Lumateperone 28 mg (ITI-007 40 mg Tosylate); Lumateperone 42 mg (ITI-007 60 mg Tosylate)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will be conducted as a randomized, double-blind, parallel-group, placebo-controlled, multi-center study in patients diagnosed with schizophrenia having an acute exacerbation of psychosis.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects of any race, ages 18-60 inclusive, with a clinical diagnosis of schizophrenia
* experiencing an acute exacerbation of psychosis

Exclusion Criteria:

* any subject unable to provide informed consent
* any female subject who is pregnant or breast-feeding
* any subject judged to be medically inappropriate for study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Vanover, Ph.D., Study Director — Intra-Cellular Therapies, Inc.
Locations (11):
- United States (11):
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Springdale, Arkansas
  - Clinical Site, Escondido, California
  - Clinical Site, Garden Grove, California
  - Clinical Site, Long Beach, California
  - Clinical Site, San Diego, California
  - Clinical Site, Fort Lauderdale, Florida
  - Clinical Site, Rockville, Maryland
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Marlton, New Jersey
  - Clinical Site, Austin, Texas

REFERENCES:
- [Derived] Citrome L, Durgam S, Edwards JB, Davis RE. Lumateperone for the Treatment of Schizophrenia: Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2023 Mar 6;84(2):22r14631. doi: 10.4088/JCP.22r14631. PMID 36883881
- [Derived] Correll CU, Davis RE, Weingart M, Saillard J, O'Gorman C, Kane JM, Lieberman JA, Tamminga CA, Mates S, Vanover KE. Efficacy and Safety of Lumateperone for Treatment of Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Apr 1;77(4):349-358. doi: 10.1001/jamapsychiatry.2019.4379. PMID 31913424

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumateperone 28 mg (ITI-007 40 mg Tosylate): Lumateperone 28 mg (ITI-007 40 mg Tosylate) administered orally as formulated capsules once daily for 28 days
  ITI-007
- Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg Tosylate) administered orally as formulated capsules once daily for 28 days
  ITI-007
- Placebo: Placebo administered orally as formulated capsules once daily for 28 days
  Placebo
Period: Overall Study
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Started | 150 | 150 | 149 (150 patients were randomized to the placebo treatment group but only 149 patients took study drug. The number completed and discontinued is based on the 149 patients that took study drug.)
Completed | 120 | 128 | 111
Not Completed | 30 | 22 | 38
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 6 | 2 | 0
Not completed — Lack of Efficacy | 11 | 6 | 17
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 8 | 10 | 16
Not completed — Other | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo | Total
Number analyzed (Participants) | 150 | 150 | 149 | 449
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (10.08) | 42.4 (10.30) | 41.4 (10.29) | 42.4 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 26 | 103
  Male | 113 | 110 | 123 | 346
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 33 | 42 | 117
  Black or African American | 94 | 108 | 96 | 298
  Asian | 6 | 1 | 1 | 8
  Other | 8 | 8 | 10 | 26
Positive and Negative Syndrome Scale (PANSS) total score [Mean (Standard Deviation); unit: units on a scale] — The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. Thus, the PANSS Total score minimum is 30 and the maximum is 210, with higher numbers indicating more severe symptoms.
  units on a scale | 89.2 (10.13) | 90.2 (9.58) | 90.6 (11.26) | 90.0 (10.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 28 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. Thus, the PANSS Total score minimum is 30 and the maximum is 210, with higher numbers indicating more severe symptoms.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Number analyzed (Participants) | 146 | 148 | 141
units on a scale | -12.9 (1.27) | -14.5 (1.25) | -10.3 (1.32)
Statistical Analysis 1: Comparison: Lumateperone 28 mg (ITI-007 40 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.182, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -2.6, 95% CI 2-sided [-6.17 to 1.05], Standard Error of Mean 1.83
Statistical Analysis 2: Comparison: Lumateperone 42 mg (ITI-007 60 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.045, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -4.2, 95% CI 2-sided [-7.75 to -0.60], Standard Error of Mean 1.82

2. Secondary Outcome: Change From Baseline to Day 28 in Clinical Global Impressions-Severity of Illness Scale
Description: The Clinical Global Impressions (CGI) Scale is a standardized assessment tool that the clinician can use to rate the severity of illness, change over time, and efficacy of medication, taking into account the subject's clinical condition and the severity of side effects. The CGI Scale consists of 3 global subscales, only one of which was used in the present study. The first subscale, Severity of Illness (CGI-S), assesses the clinician's impression of the subject's current illness state; it is often used both before and after treatment. Scores on the Severity of Illness subscale range from 1 = "not ill" at all to 7 = "among the most extremely ill."
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Number analyzed (Participants) | 146 | 148 | 141
units on a scale | -0.8 (0.08) | -0.8 (0.07) | -0.5 (0.08)
Statistical Analysis 1: Comparison: Lumateperone 42 mg (ITI-007 60 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.045, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.54 to -0.12]

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~49 days), including 28 days of double-blind treatment
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150 | 1/149
Serious Adverse Events (participants affected / at risk) | 1/150 | 0/150 | 1/149
Other Adverse Events (participants affected / at risk) | 55/150 | 70/150 | 41/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 28 mg (ITI-007 40 mg Tosylate) (N=150) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=150) | Placebo (N=149)
Convulsion (Nervous system disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 28 mg (ITI-007 40 mg Tosylate) (N=150) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=150) | Placebo (N=149)
Headache (Nervous system disorders) | 24 | 29 | 22
Somnolence (Nervous system disorders) | 17 | 26 | 6
Sedation (Nervous system disorders) | 14 | 19 | 8
Nausea (Gastrointestinal disorders) | 7 | 16 | 11
Dry Mouth (Gastrointestinal disorders) | 9 | 11 | 7
Dizziness (Nervous system disorders) | 7 | 10 | 6
Constipation (Gastrointestinal disorders) | 6 | 10 | 4
Fatigue (Nervous system disorders) | 7 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes